CLINICAL TRIAL: NCT00631267
Title: Colles Fractures, Determining the Norm in Closed Reduction Techniques
Brief Title: CoNCReTe-trial: Colles Fractures, Determining the Norm in Closed Reduction Techniques
Acronym: CoNCReTe
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to poor patient accrual
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Drs K.Kolkman, Rijnstate hospital, arnhem
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTC-502-141207
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Colles' Fracture
Keywords: reduction; satisfaction; visual-analog scale; complications; functional outcome; radiological outcome
MeSH Terms: conditions — Colles' Fracture; Personal Satisfaction | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Manual Manipulation
  Interventions: Procedure: Manual Manipulation
- 2 (Active Comparator): Finger Trap Traction
  Interventions: Procedure: Finger Trap Traction

INTERVENTIONS:
Procedure: Manual Manipulation — The currently used method for reduction: using manual traction to reduce the distal radial fragment by hyperextension followed by hyperflection.
  Arms: 1
Procedure: Finger Trap Traction — Using a finger trap traction device in vertical suspension. After 10min reduction by dorsal pressure.
  Arms: 2

SUMMARY:
Rationale:

Many different closed techniques are used to reduce a dorsally dislocated distal radius fracture (Colles' fracture). One trial to compare two main techniques (finger-trap traction and manual manipulation) did not find significant difference in radiological and clinical outcome (Earnshaw 2002). This trial aims to investigate patient and medical satisfaction between both techniques

Objective:

To demonstrate patient satisfaction (pain, duration, general) and medical satisfaction (difficulty of reposition). It is suggested that finger-trap traction causes less pain for patients and is more easy than manual manipulation but have the same radiological and clinical outcome.

Study design:

Randomised controlled intervention study

Study population:

300 Patients with newly diagnosed closed distal radius fractures with dorsal angulation (Colles' fracture) older than 16years coming to the Emergency Medical Department.

Intervention:

One group is put in finger-trap traction (digitus 1-3) for 10minutes with 4-5kg of ballast on their upper arm followed by reduction by dorsal pressure. The other group is manually reduced according to Charnley with traction and "hooking over" of the fracture elements.

Main study parameters/endpoints:

Visual analogue scale of patient and medical satisfaction, percentage of successful primary reductions. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Apart for the regular follow-up of patients with distal radius fractures,one extra out-patient visit is necessary to assess functional outcome after three months.Finger-trap traction has a (theoretical) risk of causing traumatic damage to ligaments of the fingers, but this risk is in our opinion not higher than in the manual manipulation. It is expected that the finger-trap traction group is more satisfied because this technique seems less traumatic than but as successful as the manual manipulation group.

ELIGIBILITY:
Inclusion Criteria:

Patients of 16 years and older visiting our EMD with newly diagnosed closed distal radius fractures:

* within 2cm of the radiocarpal joint
* with dorsoradial dislocation (Colles' fractures),
* AO-type 23.A2 and 23.A3 (extra-articular) and 23-C1 and 23-C2 (intra-articular)
* which are in need for reduction. I.e. Colles' fractures:

  * with loss of ≥2mm of radial height (RH),
  * change of ≥5º of radial inclination (RI),
  * loss of ≥10º volar tilt (VT),
  * loss of reduction of the distal radioulnar (DRU) joint and/or
  * fractures with >1mm intra-articular step-off

Exclusion Criteria:

* Patients who will not have their follow-up in our hospital
* Patients <16 year old
* Greenstick fractures
* Additional fractures of carpalia or elbow joint
* Patients suffering a High Energy Trauma (HET)
* Fractures that do not need reduction (see 4.2 for definition)
* Patients with pre-existent wrist-trauma or pathological bone except for osteoporosis (cyst, metastasis)
* Patients who cannot give informed consent or do not understand the Dutch language
* Patients with bilateral fractures
* Open fractures
* Fractures >48h old
* (Smith, Barton, reversed Barton or Chauffeurs fractures)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2008-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To determine the difference in satisfaction of both patient and treating doctor between two well-known techniques of fracture reposition provided that both techniques show equal results in clinical and radiological outcome. | 3 months

SECONDARY OUTCOMES:
To describe the functional outcome after three months, complication rate and osteoporosis rate in an urban community of a level-2 trauma-centre. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Karel Kolkman, MD, surgeon, Study Director — Rijnstate Hospital Arnhem
Locations (1):
- Alysis Rijnstate Hospital, Arnhem, Gelderland, Netherlands

REFERENCES:
- [Background] Earnshaw SA, Aladin A, Surendran S, Moran CG. Closed reduction of colles fractures: comparison of manual manipulation and finger-trap traction: a prospective, randomized study. J Bone Joint Surg Am. 2002 Mar;84(3):354-8. doi: 10.2106/00004623-200203000-00004. PMID 11886903